CLINICAL TRIAL: NCT03471208
Title: Dynamic Navigation-Assisted Dental Implant Placement: A Randomised Controlled Clinical Trial Comparing Accuracy With the Freehand
Brief Title: Dynamic Navigation-Assisted Dental Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Volkan Arisan, Dr. Volkan Arısan, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Navigation
Record Dates: First submitted 2018-02-22; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Dental Implants, Surgery, Computers

STUDY DESIGN:
Intervention Model Description: Dental implant surgery assisted by a stereotaxic surgical instrument
Who Masked: Investigator
Masking Description: Investigation of the post-op images included anonymized patient names providing unbiased analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dynamic Navigation (Experimental): Dental implant surgery via dynamic navigation assistance
  Interventions: Device: Dynamic Navigation Assisted Implant Surgery
- Freehand (Active Comparator): Dental implant surgery via conventional freehand
  Interventions: Procedure: Freehand Implant Surgery

INTERVENTIONS:
Device: Dynamic Navigation Assisted Implant Surgery — Implant surgery using dynamic navigation assistance
  Arms: Dynamic Navigation
Procedure: Freehand Implant Surgery — Dental implant surgery via conventional freehand
  Other Names: Dental implant surgery via conventional freehand
  Arms: Freehand

SUMMARY:
Placement of dental implants via the freehand approach may result in damage to the surrounding critical anatomy of undiscordant prosthetic position. A real-time navigational stereotaxic surgical instrument (navigation) may help to alleviate these undesired outcomes in the freehand approach.

All patients received implants in the right and left the side of their upper jaws via the random use of the navigation or the freehand approach. Positional deviations between the planned and placed implants were measured on a final tomographic image matched to the baseline.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged >18 years.
* Patients approving to participate in the trial and giving written consent
* must be able to open his/her mouth

Exclusion Criteria:

* Hemodynamically significant mitral valve stenosis
* Prosthetic heart valve (annuloplasty with or without prosthetic ring, commissurotomy and/or valvuloplasty are permitted)
* Planned cardioversion (electrical or pharmacological)
* Transient atrial fibrillation caused by a reversible disorder (e.g., thyrotoxicosis, pulmonary embolism, recent surgery, myocardial infacrtion)
* Known presence of atrial myxoma or left ventricular thrombus
* Active endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change between the planned and placed implant positions | 12 weeks
  Deviations between the planned and placed implants will be measured by matching the pre- and post-op tomographic images.

SECONDARY OUTCOMES:
Damage to the surrounding critical anatomy | 1 day (On the day of surgery).
  Any damage to the sinus maxillaries

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aydemir CA, Arisan V. Accuracy of dental implant placement via dynamic navigation or the freehand method: A split-mouth randomized controlled clinical trial. Clin Oral Implants Res. 2020 Mar;31(3):255-263. doi: 10.1111/clr.13563. Epub 2019 Dec 29. PMID 31829457